CLINICAL TRIAL: NCT01033721
Title: A Phase I Open-Label Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of Single Intravitreal and Subconjunctival Doses of Palomid 529 in Patients With Advanced Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Phase I Study of Palomid 529 a Dual TORC1/2 Inhibitor of the PI3K/Akt/mTOR Pathway for Advanced Neovascular Age-Related Macular Degeneration
Acronym: P52901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paloma Pharmaceuticals, Inc. (Industry)
Responsible Party: David Sherris, Paloma Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Paloma P529 Ocular
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — palomid 529

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Palomid 529 — comparison of different dosages of drug
  Other Names: P529

SUMMARY:
Palomid 529 is a dual TORC1/2 inhibitor of the PI3K/Akt/mTOR pathway having broad activity in angiogenesis and cellular proliferation. Palomid 529 will be examined to determine if the safety, tolerability and pharmacokinetic profile of single ascending doses when administered intravitreally or subconjunctivally.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity in the study eye between 20/100 and 20/800 (between 53 and 4 ETDRS letters read), and better or equal to 20/200 (minimum of 34 letters read) in the fellow eye.
* Subfoveal choroidal neovascularization (CNV) due to AMD
* Total area of the lesion (including blood, neovascularization and scar/atrophy) must be < 12 DA.
* Only 1 eye will be treated in the study. If both eyes are eligible, the investigator will select the eye with the most active CNV
* Clear ocular media and adequate pupillary dilatation to permit good stereo fundus photography for screening
* Intraocular pressure of 21 mm Hg or less
* Retinal thickness ≥ 250 μm by OCT, with presence of intraretinal or subretinal fluid

Exclusion Criteria:

* Any retinovascular disease or retinal degeneration other than AMD
* Serous pigment epithelial detachment without the presence of neovascularization
* Previous posterior vitrectomy or retinal surgery
* Any periocular infection in the past 4 weeks
* Concomitant therapy with anti-VEGF therapies, e.g. Avastin, Lucentis or Macugen, or previous use of these agents within 60 days of screening
* Concomitant therapy with intravenous or intravitreous corticosteroids or use within 90 days of screening
* Significant media opacities, including cataract, which might interfere with visual acuity, assessment of toxicity, or fundus photography
* Cataract surgery in the study eye within 3 months of screening
* Intraocular surgery in the study eye within 3 months of screening
* Presence of ocular infection in the study eye
* Presence of severe myopia (-8 diopters or greater) in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety-Review AEs, concomitant meds-Vitals, HR, systolic/diastolic BP, temperature, weight-ECG changes; Physical exam-Laboratory parameters-Ophthalmic exam-visual acuity, IOP, slit lamp fundus exam, fundus photography, fluorescein angiography, OCT | 43 days

SECONDARY OUTCOMES:
Efficacy-Mean change in visual acuity by ETDRS testing-Decreased leakage and/or size on FA, decreased retinal thickness in OCT-Decreased fibrosis if detectable based on fundus examination, photography, angiography and OCT | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Heier, M.D., Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lewis GP, Chapin EA, Byun J, Luna G, Sherris D, Fisher SK. Muller cell reactivity and photoreceptor cell death are reduced after experimental retinal detachment using an inhibitor of the Akt/mTOR pathway. Invest Ophthalmol Vis Sci. 2009 Sep;50(9):4429-35. doi: 10.1167/iovs.09-3445. Epub 2009 Apr 15. PMID 19369237